CLINICAL TRIAL: NCT07006987
Title: Clinical Study for HerResolve™ in Detecting the Presence of Endometriosis Among Symptomatic Women of Ages 18-49 Years Considering Laparoscopy
Brief Title: HerResolve™ in Detecting the Presence of Endometriosis Among Symptomatic Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025.270
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: To demonstrate the performance of the non-invasive blood-based test in detecting endometriosis as compared to diagnostic laparoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A non-invasive blood-based test (Experimental): A non-invasive blood-based test to detect endometriosis as compared to diagnostic laparoscopy
  Interventions: Device: A non-invasive blood-based (HerResolve)

INTERVENTIONS:
Device: A non-invasive blood-based (HerResolve) — A non-invasive blood-based test can detect endometriosis as compared to diagnostic laparoscopy

SUMMARY:
Endometriosis (EMS) is a common gynecological disease that affects 176 million girls and women globally. EMS affects 5-10% of women and adolescents within the reproductive age range of 15-49 years, and for those facing infertility, this figure may climb up to 50%. EMS can start at the first menstrual period and last until menopause. Shockingly, between 50% and 80% of women grappling with pelvic pain are found to have EMS. The formation of scar tissue (adhesions, fibrosis) within the pelvis and other parts of the body can cause severe pain and lead to infertility.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 49 with mild to severe symptoms of pelvic pain and/or abnormal bleeding.
* Diagnostic laparoscopy is scheduled with histology on any visually suspected endometriosis, and all reports (surgical and pathology) to confirm a positive result. If no visually suspicious endometriotic lesions are seen, biopsies from random areas during the laparoscopy procedure to confirm a negative histopathology result.
* Blood drawn during secretory or proliferative phase of the menstrual cycle
* Provide written informed consent to participate in the study and provide medical history on medications.

Exclusion Criteria:

* Patients who object to medical history collection and data requests
* Patients with cancer and/or undergoing chemotherapy and/or radiotherapy
* Patients who are unable or do not undergo laparoscopic surgery
* Patients participating in additional interventional clinical studies
* Pregnant, lactating, or subjects who are not healthy enough for blood donation.
* Blood drawn during menses or ovulation phase of menstrual cycle
* Females who are post-menopausa

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2037-06-01 (Estimated)

PRIMARY OUTCOMES:
Detecting endometriosis as compared to diagnostic laparoscopy | 1 week
  To demonstrate the performance of the non-invasive blood-based test in detecting endometriosis as compared to diagnostic laparoscopy

SECONDARY OUTCOMES:
Performance Objective: | 1 year
  Sensitivity: 90% (95% CI: 85%, 98%) Specificity: 90% (95% CI: 85%, 94%) Statistical Analysis will also include PPV and NPV. Sub-group analysis will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gynaecology The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided